CLINICAL TRIAL: NCT05290922
Title: The Accuracy of Host DNA CDO1 and CELF4 Methylation for Endometrial Cancer Screening: a Multi-center, Double-blind, Parallel Controlled Clinical Trials
Brief Title: DNA CDO1 and CELF4 Methylation for Endometrial Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); The Third Xiangya Hospital of Central South University (Other); Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EC-METHY3
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Endometrial Cancer; Cancer Screening; DNA Methylation; Testing Accuracy; Cervical Cytology
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Host DNA CDO1 and CELF4 methylation testing in cervical cytology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DNA methylation testing — The cervical cytology of 3 ml will be collected for the detection of DNA CDO1 and CELF4 methylation.

SUMMARY:
Based on the previous study of NCT04651738, we performed this trial to further confirm the accuracy of host DNA CDO1 and CELF4 methylation for endometrial cancer screening. This study would provide profound basis for the approval of assay kit of DNA methylation in China for endometrial screening. Four hospitals, including Peking Union Medical College Hospital, would enroll eligible patients in this study. The cervical cytology of 3 ml will be collected for the detection of DNA CDO1 and CELF4 methylation, and the results will compared with the endometrial histological pathology, which is achieved after collection of cervical cytology, by surgeries including hysteroscopy, dilation and curettage, total hysterectomy and others. The methylation testing would be double-blinded in operators and analysts. The study will enroll at least 7150 patients.

ELIGIBILITY:
Inclusion Criteria:

* With uerine and uterine cervix intact
* Aged 18 years or older
* With accessible histological results of endometrium
* Signed an approved informed consents
* With accessible cervical cytology before harvesting endometrial histology

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All participants will accept surgeries harvesting endometrial histology.
Sampling Method: Non-Probability Sample
Enrollment: 7150 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-09-12 (Estimated); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of methylation testing | One week
  Sensitivity of methylation testing of cervical cytology compared with histology
Specificity of methylation testing | One week
  Specificity of methylation testing of cervical cytology compared with histology

SECONDARY OUTCOMES:
Positive predictive value of methylation testing | One week
  Positive predictive value of methylation testing of cervical cytology compared with histology
Negative predictive value of methylation testing | One week
  Negative predictive value of methylation testing of cervical cytology compared with histology

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China